CLINICAL TRIAL: NCT06385899
Title: The Effect of Close and Intensive Therapeutic Monitoring of Patients With Poorly Controlled Type 2 Diabetes With Different Glycemic Background
Brief Title: Effect of Intensive Monitoring of Patients With Poorly Controlled Type 2 Diabetes With Different Glycemic Background
Status: Completed | Type: Observational
Sponsor: Goztepe Prof Dr Suleyman Yalcın City Hospital (Other)
Responsible Party: Principal Investigator, Ayse N Erbakan, The Principal Investigator, Goztepe Prof Dr Suleyman Yalcın City Hospital
Other Study IDs: : Poorly controlled T2DM-12
Record Dates: First submitted 2024-04-18; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Type 2 Diabetes; Poor Glycemic Control
Keywords: type 2 diabetes; poorly metabolic control
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Newly diagnosed diabetes: Patients who have been diagnosed with type 2 diabetes within a month
- Had controlled diabetes before: Patients who had at least two HbA1c levels =<%7,5 before enrollment
- Had moderately uncontrolled diabetes: Patients who had at least two HbA1c levels between %7,5 and %9,49 before enrollment
- Had poorly controlled diabetes: Patients who had at least two HbA1c levels above %9,5 before enrollment

SUMMARY:
In Turkey, only 55% of patients with type 2 diabetes have been diagnosed, and 91% of these patients have been receiving treatment. The rate of patients reaching the treatment target is 50%. The pandemic has also affected diabetic patients. It is aimed to determine the characteristics of patients with type 2 diabetes (HbA1c >=10) with poor metabolic control and to evaluate the extent to which metabolic control can be achieved in 12 months.

DETAILED DESCRIPTION:
Patients who applied to Istanbul Medeniyet University Goztepe Prof. Dr. Suleyman Yalcin City Hospital Diabetes Polyclinics and have an HbA1c levels of >= 10% in their examinations will be admitted to the study. Detailed history, including medication usage and previous blood tests will be questioned. The patients will be asked to complete questionnaires about their eating patterns (mindful eating questionnaire), their physical activities (General practice physical activity questionnaire), and whether the participants have depression (Beck depression questionnaire). Anthropometric measurements will be taken, and biochemical data will be recorded. Patients will be grouped according to their previous HbA1c values as a) newly diagnosed, b) those whose diabetes was previously controlled, c) those whose diabetes was previously not at the target range but now worsened, and d) those whose diabetes was poorly controlled from the beginning. Diabetes follow-up will be continued by their respective physicians. The patients will be called again three months after their enrollment to record the most recent biochemical data. Patient characteristics (age, gender, educational status, depression status, eating awareness, exercise characteristics) will be evaluated in accordance with the predetermined HbA1c groups. Again, according to the patient groups, the difference in HbA1c after three months, the frequency of reaching the target, and possible factors associated with the findings will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with type 2 diabetes
* give consent to the study
* accessibility to the previous and recent test results

Exclusion Criteria:

* acute infection or inflammation lasting more than a week
* acute metabolic decompensation
* unable to attend to the follow-ups
* having non-thyroid endocrine diseases
* active oncologic treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been diagnosed
Sampling Method: Non-Probability Sample
Enrollment: 266 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Changes in HbA1c levels after 12 months treatment | twelve months
  Changes in HbA1c levels after 12 months treatment according to the predetermined HbA1c groups.
percentage of patients who reached the HbA1c target of equal to or below 7% | twelve months
  Comparison of the patient groups in their success in reaching the HbA1c target of equal to or below 7%

SECONDARY OUTCOMES:
The effect of education on the HbA1c changes | twelve months
  Educational status may have an impact on HbA1c reduction. Participants who have reached the HbA1c target are compared in terms of their educational level and those who have not.
The effect of depression on the HbA1c changes | twelve months
  The Beck Depression Index will be used to compare participants who reach the HbA1c target and those who do not
The effect of the level of physical activity on the HbA1c changes | twelve months
  Physical activity is graded into 4 levels. Levels will be compared in participants who reach target HbA1c level and who do not
The effect of weight loss on the HbA1c changes | twelve months
  The effect of weight loss on reaching HbA1c target of 7% will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Ayse N Erbakan, Principal Investigator — Goztepe Prof Dr Suleyman Yalcın City Hospital
Locations (1):
- Istanbul Goztepe Prof. Dr. Suleyman Yalcin City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No